CLINICAL TRIAL: NCT00005622
Title: Allogeneic Bone Marrow Transplantation Using Closely Matched Related and Unrelated Donors
Brief Title: Donor Bone Marrow Transplant in Treating Patients With Leukemia, Lymphoma, or Nonmalignant Hematologic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11282; IRB-4189 (Other: University of South Florida IRB); NCI-G00-1755 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Multiple Myeloma and Malignant Plasma Cell Neoplasms; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute lymphoblastic leukemia; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Multiple Myeloma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cy/TBI (Other): cyclophosphamide and total body irradiation (TBI)
  Interventions: Drug: cyclophosphamide; Radiation: TBI

INTERVENTIONS:
Drug: cyclophosphamide — Cyclophosphamide is administered at a dose of 60 mg/kg on each of two successive days (Days -6 and -5)
Radiation: TBI — FTBI is performed on day -3 through day 0 The total dose of radiation is 1,320 cGy.

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related or unrelated donor, that closely matches the patient's blood, are infused into the patient they may help the patient's bone marrow to make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well donor bone marrow transplant works in treating patients with leukemia, lymphoma, or nonmalignant hematologic disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival of allogeneic bone marrow transplantation using closely matched related and unrelated donors in patients with malignant or nonmalignant hematological disorders.
* Determine the incidence and severity of acute and chronic graft versus host disease with this treatment regimen in these patients.
* Determine the relapse rates with this treatment regimen in those patients with malignant disorders.
* Determine the incidence and severity of infectious complications associated with this treatment regimen in these patients.

OUTLINE: Patients receive cyclophosphamide IV over 1 hour on days -6 and -5, total body radiotherapy on days -3 through 0, and allogeneic bone marrow transplantation on day 0.

Patients with acute lymphocytic leukemia (ALL) receive intrathecal methotrexate at the beginning of the study. If CNS involvement is documented, patients receive a second dose of methotrexate 48 hours later followed by oral leucovorin calcium every 6 hours for 4 doses. Patients with ALL and/or CNS involvement receive intrathecal methotrexate every other week for 12 weeks after transplant.

Patients with prior CNS involvement receive radiotherapy for 2.5 weeks prior to transplant. Patients with ALL receive total body radiotherapy for 5 consecutive days prior to transplant.

Patients are followed once a week for 3 months, and then monthly for 1 year.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Acute lymphocytic leukemia (ALL):

    * Complete remission (CR) 1 - high risk defined as overt CNS involvement or poor cytogenetics (additions, deletions, translocations, or multiple abnormalities)
    * CR2
    * Induction failures
    * Relapse - patients with at least 10% marrow blasts undergo at least one reinduction attempt
  * Acute myelogenous leukemia (AML):

    * CR1 - high risk defined as poor cytogenetics (deletions, additions, multiple abnormalities)
    * CR2
    * Induction failures
    * Relapse - patients with at least 10% marrow blasts undergo at least one reinduction attempt
  * Chronic myelogenous leukemia (CML):

    * Chronic phase (CP) 1
    * Accelerated phase/CP2 - patients in blast phase must undergo treatment and achieve a second chronic phase prior to transplant
  * Chronic lymphocytic leukemia (CLL):

    * Relapse - any stage; must have received no more than 3 prior regimens
  * Multiple myeloma:

    * At diagnosis - primary refractory
    * Relapse (no more than 2) - sensitive disease
    * Plasma cell leukemia
    * Inability to achieve a complete remission after autologous transplant (no older than 40)
  * Myelodysplasia - all subtypes
  * Myeloproliferative disorders - patients with poor response to medical therapy or cytogenetic abnormalities
  * Severe aplastic anemia (SAA):

    * Very SAA - at diagnosis
    * SAA - induction therapy
* Donors must be a phenotypic (6 out of 6) match or a one antigen (A or B) mismatch

PATIENT CHARACTERISTICS:

Age:

* 15 to 50

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT and SGPT no greater than 3 times normal
* PT/PTT normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* Left ventricular ejection fraction at least 45%
* No myocardial infarction within past 6 months
* No uncontrolled arrhythmias

Pulmonary:

* FEV1 at least 50%
* DLCO at least 50% predicted

Other:

* No active serious infection
* HIV negative
* Not pregnant or nursing
* No uncontrolled diabetes mellitus or thyroid disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 1996-05; Primary Completion 2005-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
event free survival (EFS) | five year post transplant
  EFS determined by the Kaplan-Meier product limit method

SECONDARY OUTCOMES:
Incidence of graft versus host disease | five years post transplant
  incidence and severity of acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Field, MD, PhD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States